CLINICAL TRIAL: NCT03016338
Title: A Phase II, Open Label Study of the Poly(ADP-ribose) Polymerase Inhibitor Niraparib in Monotherapy or in Combination With Anti-PD1 Inhibitor TSR-042 in Recurrent Endometrial Cancer
Brief Title: Study of Niraparib and TSR-042 in Recurrent Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEC
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — niraparib; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niraparib +TSR-042 (Experimental): 200/300 mg Niraparib by mouth once a day for 21 days cycle. 500 mg of TSR-042 intravenously on the first day of each cycle.
  Interventions: Drug: Niraparib; Drug: TSR-042

INTERVENTIONS:
Drug: Niraparib — 200 or 300 mg daily PO, for 21 day cycle
  Other Names: MK4827
Drug: TSR-042 — 500 mg once intravenously on day 1 of cycle (From cycle 1-4 followed by 1000 mg intravenously every 6 weeks for maximum of 2 yrs)
  Other Names: Dostarlimab

SUMMARY:
This is a phase 2 study of investigational drug niraparib and TSR-042 in patients with advanced/recurrent endometrial cancer. The purpose of this study is to determine whether blocking a protein called poly (ADP-ribose) polymerase (PARP) with niraparib provides clinical benefit in patients with recurrent endometrial cancer, as well as to explore the possible impact of phosphatase and tensin homolog (PTEN) loss (loss of function of the PTEN gene) on blocking PARP with niraparib.

DETAILED DESCRIPTION:
The purpose of this trial is to elucidate whether the PARP inhibition approach with niraparib, or the combination of niraparib and TSR-042, provides clinical benefit in patients with recurrent endometrial cancer.

The trial is designed as a multicenter, open-label, phase II study of niraparib in monotherapy or in combination with anti-PD1 inhibitor TSR-042 in recurrent endometrial cancer. Patients must have received prior platinum based chemotherapy.

The study will initially enroll patients with recurrent endometrial cancer to the niraparib monotherapy cohort not selected according to the PTEN status (cohort I).

Once the initial assessment with niraparib monotherapy is completed (inclusion of 22 evaluable patients),Additional 22 patients will be enrolled in the combination arm with niraparib and TSR-042 (cohort II).

Eligible participants will take niraparib capsules or tablets by mouth 300/200 mg, once a day, every day of every 21 day cycle.Participant will receive TSR-042 500 mg( intravenously) on the first day of each cycle for cycle 1 to 4. Followed by 1000 mg every 2 cycle for every 6 weeks for maximum of 2 yrs.

While receiving the study treatment, participants will be asked to visit the study site on Days 1, 8, 15 of Cycle 1.Cycle 2 onward Days 1 and 15 and future cycles for safety tests and procedures. If, at any time, participants develop (or is suspected to have developed) MDS/AML, a mandatory bone marrow aspirate/biopsy will be done for testing to confirm diagnosis.

When participants are taken off the study treatment permanently, they will be asked to return to the study site for an End of Study Treatment visit to have tests and procedures done for safety purposes.

Participants who are taken off the study treatment for any reason other than disease progression will continue to have radiological assessments every 8 weeks until disease progression. Participants will continue to be followed up for side effects weekly in the first 4 weeks, then monthly until resolution.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial endometrial cancer. All histological subtypes are allowed except for endometrial sarcoma, carcinosarcoma, clear cell, mixed and adenosquamous tumors.
* Patients must have radiographic evidence of disease progression following the most recent line of treatment.
* Patients must have previously received at least one line of platinum-based chemotherapy. Prior hormonal and immunotherapy are allowed. There is no restriction on the total number prior lines of therapy.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥10 mm with CT scan, MRI, or calipers by clinical exam, and ≥15mm for nodal lesions. Areas of previous radiation may not serve as measurable disease unless there is evidence of progression post radiation.
* Patients must have archival tumor sample available for PTEN analysis. If archival tissue is not available, the patient will have the option to undergo tumor biopsy.
* Eastern Cooperative Group (ECOG) performance status ≤ 2.
* Life expectancy of greater than 12 weeks.
* Within 7 days of the proposed start of treatment, patients must have normal organ and marrow function.
* Participant receiving corticosteroids may continue as long as their dose is stable for at least 4 weeks prior to initiating protocol therapy
* Patient must agree to not donate blood during the study or for 90 days after the last dose of study treatment

Exclusion Criteria:

* Chemotherapy or biologic agents received within 4 weeks of starting study treatment.
* Hormonal therapy within 2 weeks of starting study treatment.
* Pelvic radiotherapy (as treatment of primary disease) within 4 weeks, or palliative radiotherapy encompassing >20% of the bone marrow within 1 week of starting study treatment.
* Previous treatment with a PARP inhibitor, or any other targeted therapy directed against the homologous recombination pathway.
* Patients who are receiving any other investigational agents.
* Ongoing ≥ Grade 2 toxicities related to prior cancer therapy, with the exceptions of alopecia, neuropathy, lymphopenia and skin depigmentation.
* Received transfusion (platelets or red blood cells) ≤4 weeks of the first dose of study treatment.
* Major surgery within 4 weeks of registration or ongoing clinically significant post-surgical complications. Study biopsy is not considered major surgery.
* Known brain metastases, except if stable for greater than 28 days following definitive treatment. The patient must have no new or progressive signs or symptoms related to the CNS disease and must be either off or taking a stable dose of corticosteroids. A scan to confirm the absence of brain metastases is not required.
* History of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML).
* History of bowel obstruction within 3 months, or other reason preventing effective oral administration of medication.
* Immunocompromised patients e.g. Human Immunodeficiency Virus (HIV) requiring treatment or active Hepatitis B or C. Prior splenectomy is allowed.
* Uncontrolled inter-current illness.
* History of other malignancy ≤ 3 years prior to registration with the exceptions of a) cone-biopsied in situ carcinoma of the cervix uteri; b) basal or squamous cell carcinoma of the skin. All second malignancies in this context should be discussed with the Principal Investigator.
* Previous treatment with anti PD-1, anti PD-L1, anti PD-L2, anti CTLA4 agents
* History of fistula, or high-risk of developing a fistula.
* Diagnosis of immunodeficiency or systemic steroid therapy or other form of immunosuppressive therapy within 7 days prior to initiating the protocol therapy.
* Known history of human immunodeficiency virus (type 1 or 2 antibodies).
* Known active hepatitis (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected).
* Active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) Replacement therapy eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of interstitial lung disease
* Received a live vaccine within 14 days of initiating protocol therapy
* History of ≥ Grade 3 immune-related AE with prior immunotherapy, with the exception of non-clinically significant lab abnormalities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine the antitumor activity according to RECIST v 1.1 | 16 weeks
  To determine the antitumor activity of single agent niraparib and of niraparib in combination with TSR-042 in women with metastatic endometrial cancer who has received prior platinum-based chemotherapy via assessment of clinical benefit rate (complete response, partial response or stable disease ≥16 weeks), according to RECIST v 1.1.

SECONDARY OUTCOMES:
Number of side effects | 5 years
  To assess the safety and tolerability of single agent niraparib and of niraparib in combination with TSR-042.
Overall response rate | 5 years
  Overall response rate (ORR) is defined as the proportion of subjects in the analysis population who have complete response (CR) or partial response (PR) at any time during the study using RECIST
Duration of response | 5 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.
Progression free survival rate | 5 years
  Progression free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. If such an event is not observed after 6 months of follow up, patients are censored.
Overall survival rate | 5 years
  Overall survival time (OS) is defined as the time of registration to the date of death by any cause. Following the treatment discontinuation visit, survival status will be collected for all patients using acceptable means including telephone contact.

CONTACTS AND LOCATIONS:
Overall Officials: Amit M Oza, M.D., Study Director — UHN - Princess Margaret Cancer Centre
Locations (7):
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Sunnybrook Research Institute, Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre - Glen Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No